CLINICAL TRIAL: NCT00449917
Title: Study of the Effects of "Visiobiane Anti-age" Dietary Supplement on Macular Pigment Optical Density, Contrast Sensibility and Visual Acuity
Brief Title: "Visiobiane Anti-age" Effects on Vision Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PiLeJe (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P11
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Macular Pigment Optical Density
Keywords: visual caracteristics; macular pigment optical density; visual acuity; contrast sensibility; lutein; docosahexaenoic acid (DHA)
MeSH Terms: interventions — Lutein; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lutein
Drug: DHA
Drug: vitamins

SUMMARY:
The purpose of this study is to determine the benefits of "Visiobiane Anti-age" dietary supplement on macular pigment optical density, contrast sensibility and visual acuity. Additionally, the study would like to evaluate seric variations of carotenoids and the total antioxydant capacity.

DETAILED DESCRIPTION:
Visiobiane study is a randomized trial of 30 participants designed to assess the effects of oral supplementation of macular xanthophylls (lutein and zeaxanthin) and omega-3 LCPUFAs for the eyes protection. The study will enroll healthy participants aged 45 to 55 years. 15 subjects will be assigned in placebo group and 15 in experimetal group (Visiobiane anti-age). They will be supplemented for 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* healthy caucasian men
* age : 45-55
* BMI < 25

Exclusion Criteria:

* non healthy
* retinian and/or visual anomaly
* Ocular media not clear enough to allow good fundus photography

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
macular pigment optical density

SECONDARY OUTCOMES:
contrast sensibility
visual acuity
seric carotenoids concentrations
total antioxidant capacity
influence of SR-B1 genetic polimorphism

CONTACTS AND LOCATIONS:
Overall Officials: Franck Bacin, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CRNH Clermont-Ferrand, Clermont-Ferrand, Auvergne, France